CLINICAL TRIAL: NCT06271460
Title: Answerability and Minimal Clinical Significance of the Turkish Versions of the Roland-Morris Disability Questionnaire, Quebec Low Back Pain Disability Scale, and Oswestry Disability Index in Patients With Non-specific Chronic Low Back Pain
Brief Title: Disability in Patients With Non-specific Chronic Low Back Pain
Status: Recruiting | Type: Observational
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-21-728
Record Dates: First submitted 2024-02-14; First posted 2024-02-21 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Chronic Nonspecific Low Back Pain
Keywords: chronic low back pain; disability; minimal clinically significant difference

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Other: Traditional physiotherapy — All participants will receive a 60-minute individual treatment program consisting of 16 sessions of routine physiotherapy aimed at reducing pain and improving function over four weeks. These treatments are already the patient's routine physiotherapy modalities. No changes will be made to the study.

SUMMARY:
To investigate the reliability and sensitivity of the Turkish versions of the Roland-Morris Disability Questionnaire, The Quebec Back Pain Disability Scale, and the Oswestry Disability Index in patients with chronic non-specific low back pain and to increase confidence in their use in clinical practice and research by determining the most appropriate minimal clinically significant difference values for this patient population.

DETAILED DESCRIPTION:
The minimum clinically important difference (MCID) for nonspecific chronic low back pain and disability scales varies depending on the questionnaire used and the method used to assess the MCID. Different surveys have been proposed in the areas of pain intensity, disability-specific to low back pain, patient satisfaction with treatment results, and work disability. Validated and widely used questionnaires for disability assessment include the Roland-Morris Disability Questionnaire (RMDQ) the Quebec Back Pain Disability Scale (QBPDS) and the Oswestry Disability Index (ODI). These scales are valuable tools for assessing the level of disability and functional limitations in individuals with nonspecific chronic low back pain and play a crucial role in monitoring patients' progress and comparing the effectiveness of different interventions.

ELIGIBILITY:
Inclusion Criteria:

* Getting diagnosed with chronic non-specific low back pain
* Being able to read and speak Turkish
* Being between the ages of 18 and 65
* Agreeing to participate in the research and signing the voluntary consent form

Exclusion Criteria:

* Presence of systemic disease
* Cognitive impairment status (Mini-Mental State Examination <24),
* Recent (<12 weeks) history of myocardial infarction, cerebrovascular accident
* Presence of radiculopathy, infection, tumor, osteoporosis, vertebral fracture, trauma and surgery in the lumbar region
* Having received any exercise therapy before
* Refusal of treatment or failure to comply with treatment

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 100 patients diagnosed with chronic nonspecific low back pain (documented history of low back pain lasting more than twelve weeks without a recognizable, specific pathoanatomical cause of the pain) who applied to the Physical Therapy and Rehabilitation Polyclinic of the hospitals in the Acıbadem Health Group and the Physiotherapy and Rehabilitation Department of Avicenna Ataşehir Hospital will be included in the study. Diagnoses will be made by Health Physical Medicine and Rehabilitation Doctors with at least 20 years of experience.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | baseline and through study completion, an average of 4 weeks
  Visual Analog Scale (VAS) is a pain rating scale used in clinical and research settings to measure the intensity or frequency of various symptoms. In the current study, VAS will be used to record participants' pain intensity. VAS consists of a single 10 cm line; The left end is described as "No pain" and the right end is described as "The most severe pain ever experienced". Patients will be asked to mark the severity of their current pain on a 10 cm line. When calculating, the marked point will be measured in cm. An increase in the score means that the intensity of the pain increases.
The Roland-Morris Disability Questionnaire | baseline and through study completion, an average of 4 weeks
  The Roland-Morris Disability Questionnaire (RMDQ) is a tool used to assess the disability of individuals with low back pain. In the current study, the RMDQ will be used to evaluate how participants' low back pain affects functional activities. The survey, which focuses on physical functions related to low back pain, consists of 24 questions. The questionnaire is most sensitive for patients with mild to moderate disability due to acute, subacute, or chronic low back pain. It is sensitive to change over time and has been shown to provide reliable measurements in determining the level of disability. The higher the score (0-24), the higher the level of pain-related disability.
The Quebec Back Pain Disability Scale | baseline and through study completion, an average of 4 weeks
  The Quebec Back Pain Disability Scale (QBPDS) is a condition-specific questionnaire designed to measure the level of functional disability of patients with low back pain. In the current study, QBPDS will be used to evaluate the disability of patients with low back pain during functional skills. The QBPDS consists of 20 items regarding daily activities selected from six relevant subdomains of functional skills for patients with low back pain. The scale is scored on a Likert scale from 0 to 5; 0 means "not difficult at all" and 5 means "I can't do it". The total score can range from 0 to 100; a higher score indicates a more severe disability. The minimum detectable change (90% confidence) for QBPDS is 15 points.
The Oswestry Disability Index | baseline and through study completion, an average of 4 weeks
  The Oswestry Disability Index (ODI) is a self-completed questionnaire used to assess the level of disability in patients with low back pain. In the current study, the ODI will be used to evaluate the impact of low back pain on patients' daily lives.The survey consists of ten sections focusing on different aspects of daily life, such as pain severity, personal care, weight lifting, walking, sitting, standing, sleep, sexual function, social life, and travel. Each section contains six statements scored from 0 to 5; The first expression is zero, indicating no disability. The scores of all questions are summed and then multiplied by two to obtain an index ranging from 0 to 100. The higher the score, the greater the disability.
The Perceived Global Impact | through study completion, an average of 4 weeks
  The Perceived Global Impact Scale is a tool used to assess the impact of various factors on an individual's health and well-being. In the current study, the amount of improvement in symptoms perceived by participants will be assessed at the end of treatment with the Perceived Global Impact Scale. Participants were asked, "How would you describe your current situation compared to the beginning of treatment?" The question was asked. questions will be asked. They will be asked to rate on a seven-point Likert scale (1: no change or things have gotten worse; 7: much better, a significant improvement). A score of 6 or above will be chosen as the threshold for clinically significant improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Elif E Safran, asst. prof., Principal Investigator — Acibadem University; Irmak I Çavuşoğlu, asst. prof., Study Chair — Acibadem University; Nuray N Alaca, assoc. prof., Study Director — Acibadem University
Locations (1):
- Acıbadem Health Group, Istanbul, None Selected, Turkey (Türkiye)